CLINICAL TRIAL: NCT06653946
Title: the Predictors of Different ECASS-based Hemorrhagic Transformation Subtypes in Acute Embolic Stroke Patients Treated With Alteplase
Brief Title: the Predictors of Hemorrhagic Transformation Subtypes in Acute Embolic Stroke Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, principal investigator, Kafrelsheikh University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010120190
Record Dates: First submitted 2024-10-04; First posted 2024-10-23 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke; Alteplase Adverse Reaction
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: The study consisted of two distinct groups. The first group comprised 454 patients who did not experience hemorrhagic infarction, while the second group comprised 252 patients who experienced hemorrhagic infarction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemorragic transformation group (Active Comparator): 262 acute ischemic stroke (AIS) patients who had a hemorrhagic transformation of brain infarction after 24-36 hours of receiving alteplase.
  Interventions: Drug: Alteplase
- non-hemorragic transformation group (Active Comparator): 454 acute ischemic stroke (AIS) patients did not have a hemorrhagic transformation of brain infarction after 24-36 hours of receiving alteplase
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — Following the guidelines set by the American Heart Association/American Stroke Association (AHA/ASA), inclusion and exclusion criteria for alteplase were established; 0.9 mg/kg of alteplase up to a maximum dose of 90 mg was administered intravenously to eligible individuals within 4.5 hours of the beginning of their clinical manifestations (10% bolus, 90% infusion in 1 hour). After receiving IV-alteplase, all patients continued their management and rehabilitation in the stroke unit
  Other Names: group A
  Arms: Hemorragic transformation group
Drug: Alteplase — Following the guidelines set by the American Heart Association/American Stroke Association (AHA/ASA), inclusion and exclusion criteria for alteplase were established; 0.9 mg/kg of alteplase up to a maximum dose of 90 mg was administered intravenously to eligible individuals within 4.5 hours of the beginning of their clinical manifestations (10% bolus, 90% infusion in 1 hour). After receiving IV-alteplase, all patients continued their management and rehabilitation in the stroke unit
  Other Names: group B
  Arms: non-hemorragic transformation group

SUMMARY:
The investigators evaluated the impact of AF on different subtypes of post-alteplase hemorrhagic transformation of brain infarction.

DETAILED DESCRIPTION:
Investigators conducted a prospective cohort study between July 2021 and July 2023. They screened 1550 patients who presented with AIS and received alteplase and included 716 AIS patients who met the inclusion criteria and were diagnosed based on a thorough clinical assessment, including a detailed medical history, physical examination, and specific brain imaging results and treated with alteplase within four and half hours of stroke onset.

The investigators assessed the patients' follow-up brain imaging to detect the subtypes of hemorrhagic transformation after receiving alteplase.

The study consisted of two distinct groups. The first group consisted of 454 patients who did not experience hemorrhagic infarction, while the second group comprised 262 patients who experienced hemorrhagic infarction.

The investigators evaluated whether the characteristics of ischemic stroke patients, door-to-needle time, and stroke risk factors different types of AF were predictive variables for different subtypes of post-alteplase hemorrhagic transformation of brain infarction.

ELIGIBILITY:
Inclusion Criteria:

* The investigators enrolled individuals of both genders, aged between 18 and 75,
* All patients had acute first-ever embolic ischemic stroke and were eligible for thrombolysis.
* All patients had Atrial fibrillation

Exclusion Criteria:

* The investigators excluded patients who had alteplase contraindications
* The investigators excluded patients who did not receive the total dose of alteplase for any reason.
* The investigators excluded patients who had a known history of persistent or recurrent CNS pathology (e.g., epilepsy, meningioma, multiple sclerosis)
* The investigators excluded patients who had recurrent ischemic stroke diagnosed by appropriate clinical history and/or MRI brain findings.
* The investigators excluded patients with symptoms of major organ failure, active malignancies, or an acute myocardial infarction within the previous six weeks.
* The investigators also excluded pregnant and lactating patients with stroke due to venous thrombosis and stroke following cardiac arrest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
the rate of each AF type in the hemorrhagic infarction type 1 group compared to non HT group | 48 days
  The investigators will evaluate the rate of each AF type in the hemorrhagic infarction type 1 group compared to non HT group

SECONDARY OUTCOMES:
the rate of each AF type in the hemorrhagic infarction type 2 group compared to non HT group | 48 hours
  The investigators will evaluate the rate of each AF type in the hemorrhagic infarction type 2 group compared to non HT group
the rate of each AF type in the parenchymal haematoma type 1 group compared to non HT group | 48 hours
  The investigators will evaluate the rate of each AF type in the parenchymal haematoma type 1 group compared to non HT group
the rate of each AF type in the parenchymal haematoma type 2 group compared to non HT group | 48 hours
  The investigators will evaluate the rate of each AF type in the parenchymal haematoma type 2 group compared to non HT group

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Principal Investigator — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data supporting this research's findings may be available from the principal investigator, Mohamed G. Zeinhom, upon reasonable request.

REFERENCES:
- [Result] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Result] Zeinhom MG, Aref HM, El-Khawas H, Roushdy TM, Shokri HM, Elbassiouny A. A pilot study of the ticagrelor role in ischemic stroke secondary prevention. Eur Neurol. 2022;85(1):50-55. doi: 10.1159/000518786. Epub 2021 Aug 30. PMID 34515113
- [Result] Bruno A, Levine SR, Frankel MR, Brott TG, Lin Y, Tilley BC, Lyden PD, Broderick JP, Kwiatkowski TG, Fineberg SE; NINDS rt-PA Stroke Study Group. Admission glucose level and clinical outcomes in the NINDS rt-PA Stroke Trial. Neurology. 2002 Sep 10;59(5):669-74. doi: 10.1212/wnl.59.5.669. PMID 12221155
- [Derived] Ahmed SR, Zeinhom MG, Ebied AAMK, Kamel IFM, Almoataz MA, Daabis AMA, Akl AZO, Mahmoud ELA, Alkhalefeh AG, Ouf SG, Mosbah SAA, Sirag IMI, Abouelnaga M, Khalil MFE. A multi-center study on the predictors of different subtypes of hemorrhagic transformation of brain infarction after thrombolysis in atrial fibrillation patients presented with embolic stroke. Sci Rep. 2025 May 5;15(1):15655. doi: 10.1038/s41598-025-97968-3. PMID 40325067